CLINICAL TRIAL: NCT03032224
Title: Analysis of Sarcopenia and Body Composition in Relation to Outcome in a Cohort of Patients With Esophageal Cancer or Cancer of the Gastroesophageal Junction Before and After Surgery With Curative Intent
Brief Title: Analysis of Body Composition in Relation to Outcome After Surgery in a Cohort of Patients With Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Sahlgrenska University Hospital (Other); The Göteborg Medical Society, Sweden (Unknown)
Responsible Party: Sponsor
Other Study IDs: janpe4
Record Dates: First submitted 2017-01-04; First posted 2017-01-26 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Cancer of Esophagus; Gastric Cancer
Keywords: Body composition; sarcopenia; Dysphagia; Surgery; Quality of Life; Morbidity
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Sarcopenia; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Resection of the esophagus and the gastroesophageal junction

SUMMARY:
The occurrence of dysphagia is a well-known early feature of esophageal cancer that may reduce caloric intake and thus cause weight loss. Sarcopenia is considered to be a consequence of such involuntary nutritional restriction. The prevalence of sarcopenia in patients with esophageal cancer before and after surgery is not well known and its possible consequences have been debated.

Aim: The aim of this study was to prospectively explore body composition and function in a cohort of patients with esophageal cancer before and after surgery with curative intent. In particular, to investigate the prevalence and development of sarcopenia and body composition as a consequence to surgery for esophageal cancer and the possible relation to morbidity, length of stay and quality of life (QoL).

Methods: In a cohort of 76 patients who had esophageal- or cardia-cancer and were planned for surgery with a curative intent, data on body-composition measured with bioimpedance, working capacity (cardiac stress test), grip strength and QoL (European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires (QLQ)-C30 version 3.0) were prospectively collected. Data regarding dysphagia was derived from an esophagus related quality of life form (EORTC QLQ-OES18). Data on tumour stage and type, complications, length of stay and preoperative weight loss were collected from medical charts.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the gastro-esophageal junction or the esophagus.
* Planned for curative surgery.
* Informed consent

Exclusion Criteria:

* Not fulfilling the above.
* Patient declined participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was a prospective collected cohort study in 76 patients who were referred to the surgery clinic at the Sahlgrenska University hospital 2005-2010. Patients with esophageal cancer or cancer of the gastroesophageal junction (Siewert I or II), who were scheduled to undergo resection surgery with curative intent, were asked to participate. Patients were excluded if they were found to have an advanced tumour stage or if they declined participation.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Changes in Body composition after surgery for esophageal cancer with curative intent. | Three months
  Body mass index (BMI) kg/m2
Changes in Body composition after surgery for esophageal cancer with curative intent | Three months
  Weight kg
Changes in Body composition after surgery for esophageal cancer with curative intent. | Three months
  Fat free mass (FFM) kg;
Changes in Body composition after surgery for esophageal cancer with curative intent. | Three months
  Fat mass (FM) kg;
Changes in Body composition after surgery for esophageal cancer with curative intent. | Three months
  Lean tissue mass (LTM) kg;
Changes in Body composition after surgery for esophageal cancer with curative intent. | Three months
  Total body water (TBW) l;
Changes in Body composition after surgery for esophageal cancer with curative intent. | Three months
  Intra cellular water (ICW) l;
Changes in Body composition after surgery for esophageal cancer with curative intent. | Three months
  Extra cellular water (ECW) l

SECONDARY OUTCOMES:
Changes in QoL (linear scale 0-100) | From surgery up to three months
Changes in dysphagia (linear scale 0-100) | From surgery up to three months
Length of stay (days) | From surgery up to three months
Complications after surgery (Clavien-Dindo scale 0-5) | From surgery up to three months
Mortality | Length of survival after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Department, Sahlgrenska University Hospital, Gothenburg, Västra Götalandsregionen, Sweden

IPD SHARING:
Plan to Share IPD: No